CLINICAL TRIAL: NCT00774488
Title: Acute Effects of Glucose Dependent Insulinotropic Polypeptide (GIP) on Subcutaneous Adipose Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: AFH. Pfeiffer, German Institute of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: GIP-Genexpression Study
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Metabolic Syndrome; Obesity; Insulin Sensitivity
Keywords: Euglycemic-hyperinsulinemic clamp; fat biopsies; microarray analysis; quantitative real time PCR; overnutrition; low grade-inflammation
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Insulin Resistance; Overnutrition | interventions — Incretins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Glucose dependent insulinotropic polypeptide (GIP) — GIP-Infusions for 4 h in a postprandial concentration

SUMMARY:
This clinical, randomized, cross-over study in obese healthy subjects aimed to analyse the acute effects of the incretin hormon Glucose Dependent Insulinotropic Polypeptide (GIP) on metabolic parameters and gene expression in subcutaneous adipose tissue.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 28
* Healthy subjects
* Normal glucose tolerance

Exclusion Criteria:

* Diabetes,IFG, IGT
* Chronical-inflammatory diseases
* Hb < 12g/dl
* Elevation in liver enzymes or creatinin concentrations
* Great weight changes within last 12 months
* Any cancer diagnosis in last 10 years

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Changes in gene expression of subcutaneous adipose tissue with microarray analysis | 3 years

SECONDARY OUTCOMES:
Analysis of inflammatory marker (blood levels and gene expression), Activity of 11beta HSD and 11-beta HSD mRNA in adipose tissue, etc. | 3 years

REFERENCES:
- [Derived] Tuvia N, Pivovarova-Ramich O, Murahovschi V, Luck S, Grudziecki A, Ost AC, Kruse M, Nikiforova VJ, Osterhoff M, Gottmann P, Gogebakan O, Sticht C, Gretz N, Schupp M, Schurmann A, Rudovich N, Pfeiffer AFH, Kramer A. Insulin Directly Regulates the Circadian Clock in Adipose Tissue. Diabetes. 2021 Sep;70(9):1985-1999. doi: 10.2337/db20-0910. Epub 2021 Jul 5. PMID 34226282
- [Derived] Gogebakan O, Osterhoff MA, Schuler R, Pivovarova O, Kruse M, Seltmann AC, Mosig AS, Rudovich N, Nauck M, Pfeiffer AF. GIP increases adipose tissue expression and blood levels of MCP-1 in humans and links high energy diets to inflammation: a randomised trial. Diabetologia. 2015 Aug;58(8):1759-68. doi: 10.1007/s00125-015-3618-4. Epub 2015 May 21. PMID 25994074
- [Derived] Rudovich N, Pivovarova O, Gogebakan O, Sparwasser A, Doehner W, Anker SD, Arafat AM, Bergmann A, Nauck MA, Pfeiffer AF. Effect of exogenous intravenous administrations of GLP-1 and/or GIP on circulating pro-atrial natriuretic peptide in subjects with different stages of glucose tolerance. Diabetes Care. 2015 Jan;38(1):e7-8. doi: 10.2337/dc14-1452. No abstract available. PMID 25538323